CLINICAL TRIAL: NCT00238641
Title: "DOES MYOBLOC™ IMPROVE FUNCTIONAL HAND USE IN YOUNG CHILDREN WITH A HYPERTONIC UPPER EXTREMITY?"
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Elan Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Myobloc2002
Record Dates: First submitted 2005-10-11; First posted 2005-10-13 (Estimated); Last update posted 2005-10-13 (Estimated); Status verified 2005-10

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — rimabotulinumtoxinB

INTERVENTIONS:
Drug: Botulinum Toxin type B

SUMMARY:
In children with cerebral palsy, stiffness of the arm can develop early and delay or prevent the acquisition of normal hand skills. Improvement in functional use of the hand may therefore be dependent upon early treatment of upper extremity hypertonia. We propose to test a series of injections of Myobloc™ in a non-randomized one-way crossover pilot clinical trial and dose-finding study, with clinical assessments and blinded video evaluations. Ten children age 2-17 years with increased tone at the elbow or wrist will be expected to complete the study. A 1-month baseline evaluation period will be followed by an injection of low-dose Myobloc™ to affected muscle(s) of the arm according to standardized per-kilogram dosing with a maximum of 25U/kg in each affected arm. Three months later, a second injection of up to 50U/kg will be performed in each affected arm. Three months after the second dose, a third dose of up to 100U/kg will be performed in each affected arm. Neurological assessments will be performed at study entry, prior to each injection, and at 1 and 3 months following each injection. Routine physical therapy and non-study medications will be continued during the study.

DETAILED DESCRIPTION:
Subjects: 10 subjects age 2-17 years with hypertonia affecting one or both upper extremities, but without injections of neuromuscular blocking agents for six months prior to enrollment, or surgery on the upper extremity.

Intervention: Injection of Myobloc™ in 2 sites per muscle for up to two muscles of each upper extremity (biceps, brachioradialis), at a maximum dose of 25Units/kg/arm for the first injection, a maximum of 50Units/kg/arm for the second injection, and a maximum of 100Units/kg/arm for the third injection. If there is significant weakness or worsening of function following any injection, the dose will not be increased for subsequent injections. Injections will be performed after placement of topical anesthetic (ELA-MAX™ cream), using EMG guidance to identify active muscles contributing to hypertonia.

Primary outcome measures: The primary outcome measure is the time it takes to complete maximum arm extension during voluntary reaching, measured from the coraco-acromial joint to the midpoint of the dorsum of the wrist. Change scores will be calculated between intake and 1 month (baseline effect), 1 month and 2 months (first injection effect), 4 months and 5 months (second injection effect), and 7 months and 8 months (third injection effect). A device called a Shape Tape (Measureand, Inc.) will be used to measure this outcome. Shape Tape is a flexible strip of portable spring steel with optic fiber that provides instantaneous readouts to a portable computer of bends and twists and other forms of movement capture that can be conducted in a clinical setting. The Shape Tape is fastened loosely to the body part under measurement (in this case, the subject's wrist and shoulder) with either medical-grade adhesive tape or Velcro. The shapetape is connected to a portable computer, and custom software allows measurement of the average velocity of hand movement during reaching.

Secondary outcome measures: The rater will compare improvement or worsening in global arm function through the Unified Dystonia Rating Scale (UDRS), the motor subscale of the Unified Parkinson's Disease rating scale (UPDRS), and the Burke-Fahn-Marsden dystonia scale (BFM). Comparisons will be performed between intake and 1 month (baseline effect), 1 month and 2 months (first injection effect), 4 months and 5 months (second injection effect), and 7 months and 8 months (third injection effect). Other secondary measures include neurological examination, Ashworth spasticity scale, and comparisons of numerical stiffness measures as measured by the Rigidity Analyzer Device. A parent rating scale, the Pediatric Quality of Life Inventory (PedsQL), will be used to determine overall functional improvement.

Statistical analysis: The outcomes will be tested at the 0.05 level of significance using repeated-measures analysis of variance (ANOVA) and the Friedman nonparametric test applied to the 4 repeated change scores for each of the primary and secondary outcome measures. Tests of significance for the secondary measures will be corrected for multiple comparisons.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 2- 17 years 2. Hypertonia affecting one or both upper extremities 3. Hypertonia caused by static encephalopathy due to prenatal or perinatal injury 4. Cognitive and motor function sufficient so that the child will reliably reach toward a target or a small toy 5. Concurrent enrollment in "standard of care" physical therapy or occupational therapy services

Exclusion Criteria:

* 1. Injection of neuromuscular blocking agents to any extremity within six months prior to enrollment 2. Dose changes of trihexyphenidyl, dantrolene, baclofen, dopaminergic agents or benzodiazepines during the course of the study.

  3. Any use of aminoglycoside antibiotics during the study. 4. Prior surgery to either upper extremity 5. Initiation or change in physical or occupational therapy regimen within 3 months of study entry 6. Progressive or neurodegenerative disease, or suspicion of an inborn error of metabolism 7. Neuropathy, myopathy, or neuromuscular junction disease 8. Congenital deformities of either upper extremity 9. Respiratory or airway compromise, or use of respiratory medications 10. Cardiomyopathy 11. Any other medical condition that would place the child at risk for participation

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10
Dates: Start 2002-01; Study Completion 2005-05

PRIMARY OUTCOMES:
The primary outcome measure is the time it takes to complete maximum arm extension during voluntary reaching, measured from the coraco-acromial joint to the midpoint of the dorsum of the wrist.

SECONDARY OUTCOMES:
The rater will compare improvement or worsening in global arm function through the Unified Dystonia Rating Scale (UDRS), the motor subscale of the Unified Parkinson's Disease rating scale (UPDRS), and the Burke-Fahn-Marsden dystonia scale (BFM). Compar

CONTACTS AND LOCATIONS:
Overall Officials: Terence Sanger, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States